CLINICAL TRIAL: NCT02047474
Title: Phase II Study of Peri-Operative Modified Folfirinox in Localized Pancreatic Cancer
Brief Title: Combination Chemotherapy Before and After Surgery in Treating Patients With Localized Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1306012255; NCI-2013-02349 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1306012255 (Other: Yale University); P30CA016359 (NIH)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Stage I Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

ARMS (1):
- Treatment (mFOLFIRINOX) (Experimental): NEOADJUVANT THERAPY: Patients receive mFOLFIRINOX comprising oxaliplatin IV over 2 hours, levoleucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV continuously for 46 hours on day 1. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  SURGERY: Beginning 3-8 weeks after completion of neoadjuvant therapy patients undergo surgical resection.
  ADJUVANT THERARPY: Beginning within 12 weeks after surgery, patients receive mFOLFIRINOX as in neoadjuvant therapy. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: irinotecan hydrochloride; Drug: fluorouracil; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well combination chemotherapy before and after surgery works in treating patients with localized pancreatic cancer. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, irinotecan hydrochloride, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival in patients with resectable non-metastatic pancreatic cancer treated with peri-operative modified leucovorin calcium, fluorouracil, irinotecan hydrochloride, oxaliplatin (mFOLFIRINOX).

SECONDARY OBJECTIVES:

I. Determine overall survival. II. Determine objective response rate after neoadjuvant mFOLFIRINOX.

TERTIARY OBJECTIVES:

I. Compare R0 resection rate and pathologic stage with institutional historical controls who did not receive neoadjuvant therapy.

II. Correlate early metabolic response, determined by changes in glucose metabolism using positron emission tomography (PET) scanning, with pathologic response, R0 resection, and pathologic stage.

III. Correlate early metabolic response, determined by changes in glucose metabolism using PET scanning, with progression-free and overall survival.

IV. Correlate pre-operative response of CA19-9 with progression-free and overall survival.

V. Collect and bank serial serum and plasma specimens from subjects for future correlative biomarker studies.

VI. Collect and bank tumor tissue from subjects prior to treatment (from the diagnostic endoscopic ultrasonography [EUS]-guided biopsy) and after treatment with six cycles of FOLFIRINOX (from the surgical specimen) for future correlative biomarker studies.

OUTLINE:

NEOADJUVANT THERAPY: Patients receive mFOLFIRINOX comprising oxaliplatin intravenously (IV) over 2 hours, levoleucovorin calcium IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and fluorouracil IV continuously for 46 hours on day 1. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

SURGERY: Beginning 3-8 weeks after completion of neoadjuvant therapy patients undergo surgical resection.

ADJUVANT THERARPY: Beginning within 12 weeks after surgery, patients receive mFOLFIRINOX as in neoadjuvant therapy. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 3 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic or cytologic documentation of pancreatic adenocarcinoma
* Resectable pancreatic adenocarcinoma disease as defined as follows:

  * No evidence of extrapancreatic disease by cross sectional imaging, PET scan, or laparoscopy, including nodal involvement beyond the peripancreatic tissues and/or distant metastases;
  * No evidence of tumor extension to superior mesenteric artery, hepatic artery, celiac axis, aorta, or inferior vena cava, and no evidence of occlusion or encasement of the superior mesenteric vein or superior mesenteric vein/portal vein confluence, as assessed by computed tomography (CT) using pancreatic protocol (or magnetic resonance imaging [MRI] in patients who cannot undergo CT) and EUS
* No prior treatment (chemotherapy, biological therapy, or radiotherapy) for resectable pancreatic cancer
* No prior treatment with oxaliplatin, irinotecan (irinotecan hydrochloride), fluorouracil or capecitabine
* Patients who received chemotherapy > 5 years ago for malignancies other than pancreatic cancer are eligible
* There is no evidence of the second malignancy at the time of study entry
* > 4 weeks since major surgery
* No other concurrent anticancer therapy
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-1
* No other malignancy within past five years except basal cell carcinoma of the skin, cervical carcinoma in situ, or non-metastatic prostate cancer
* Paraffin block or slides must be available
* Adequate organ function
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No >= grade 2 sensory peripheral neuropathy
* No uncontrolled seizure disorder, active neurological disease, or known central nervous system (CNS) disease
* No significant cardiac disease, including the following: unstable angina, New York Heart Association class II-IV congestive heart failure, myocardial infarction within six months prior to study enrollment
* No history of chronic diarrhea
* Not pregnant and not nursing
* No other medical condition or reason that, in the opinion of the investigator, would preclude study participation
* Absolute neutrophil count >= 1,500/uL
* Platelet count >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Creatinine < 1.5 X upper limit of normal (ULN) or
* Estimated glomerular filtration rate (GFR) > 30 ml/min
* Bilirubin =< 1.5 X ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 X ULN
* Negative pregnancy test in women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate | At 12 months
  Evaluated using a one-sided 0.10-alpha level exact test. Summarized using Kaplan-Meier curves

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  Summarized using Kaplan-Meier curves.
Objective response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jill Lacy, MD, Principal Investigator — Yale University
Locations (9):
- United States (9):
  - Smilow Cancer Hospital at Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital at Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital at St. Francis Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital at North Haven, North Haven, Connecticut
  - Smilow Cancer Hospital at Orange, Orange, Connecticut
  - Smilow Cancer Hospital at Torrington, Torrington, Connecticut
  - Smilow Cancer Hospital at Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital at Waterbury, Waterbury, Connecticut

REFERENCES:
- [Derived] Cecchini M, Salem RR, Robert M, Czerniak S, Blaha O, Zelterman D, Rajaei M, Townsend JP, Cai G, Chowdhury S, Yugawa D, Tseng R, Mejia Arbelaez C, Jiao J, Shroyer K, Thumar J, Kortmansky J, Zaheer W, Fischbach N, Persico J, Stein S, Khan SA, Cha C, Billingsley KG, Kunstman JW, Johung KL, Wiess C, Muzumdar MD, Spickard E, Aushev VN, Laliotis G, Jurdi A, Liu MC, Escobar-Hoyos L, Lacy J. Perioperative Modified FOLFIRINOX for Resectable Pancreatic Cancer: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Aug 1;10(8):1027-1035. doi: 10.1001/jamaoncol.2024.1575. PMID 38900452